CLINICAL TRIAL: NCT02854813
Title: Overactive Bladder in Elderly Patients- An Early Warning of Coronary Artery Disease
Status: Completed | Type: Observational
Sponsor: Ankara Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Muhammet Fatih Kilinc, M.D., Ankara Training and Research Hospital
Other Study IDs: 5192
Record Dates: First submitted 2016-07-31; First posted 2016-08-03 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Overactive Bladder Syndrome; Coronary Artery Disease
Keywords: overactive bladder; coronary artery disease; gensini score
MeSH Terms: conditions — Coronary Artery Disease; Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: Patients with a OAB-V8 score ≥8
- Group 2: Patients with a OAB-V8 score <8

SUMMARY:
Investigators aimed to investigate the association between over active bladder and coronary artery disease as demonstrated on coronary angiography.

DETAILED DESCRIPTION:
The close relationship has been demonstrated between pelvic ischemia and overactive bladder (OAB) in a study involving elderly patients. In this study, it has been found that pelvic ischemia has triggered OAB and it has been related with cardiac ischemia. The aim of this study was to delineate the correlation between OAB and the degree of coronary artery stenosis as demonstrated on coronary angiography.

ELIGIBILITY:
Inclusion Criteria:

* patients, whom were diagnosed to undergo coronary angiography in a center of cardiology

Exclusion Criteria:

* a maximum flow rate of 15 ml. per second or less,
* residual volume of 100 cc or more,
* diabetes mellitus,
* neurologic disease,
* prostate or bladder cancer,
* renal failure,
* urinary tract infection,
* nephrolithiasis or pelvic surgery,
* patients with a history of percutaneous coronary intervention or coronary artery bypass grafting

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: patients, whom were diagnosed to undergo coronary angiography in a center of cardiology between January 2016 and January 2017 were evaluated prospectively.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2016-01; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Over active bladder V8 questionnaire score | 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Tarcan T, Azadzoi KM, Siroky MB, Goldstein I, Krane RJ. Age-related erectile and voiding dysfunction: the role of arterial insufficiency. Br J Urol. 1998 Dec;82 Suppl 1:26-33. doi: 10.1046/j.1464-410x.1998.0820s1026.x. No abstract available. PMID 9883259
- [Background] De EJ, Hou P, Estrera AL, Sdringola S, Kramer LA, Graves DE, Westney OL. Pelvic ischemia is measurable and symptomatic in patients with coronary artery disease: a novel application of dynamic contrast-enhanced magnetic resonance imaging. J Sex Med. 2008 Nov;5(11):2635-45. doi: 10.1111/j.1743-6109.2008.00969.x. Epub 2008 Aug 26. PMID 18761598